CLINICAL TRIAL: NCT01076257
Title: Efficacy of Modified Constraint-induced Movement Therapy in Children With Brain Damage: Evidence of Kinematic Study
Brief Title: Efficacy of Modified Constraint-induced Movement Therapy in Children With Brain Damage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 97-1823B
Record Dates: First submitted 2010-01-04; First posted 2010-02-26 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2010-05

CONDITIONS: Brain Damage; Cerebral Palsy; Traumatic Brain Damage
Keywords: brain damage; constraint induced movement therapy; kinematic; function; outcome; Quality of life
MeSH Terms: conditions — Brain Injuries; Cerebral Palsy; Brain Injuries, Traumatic | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Constraint-induced Movement Therapy (Experimental)
  Interventions: Behavioral: Modified Constraint-induced Movement Therapy
- Transditional rehabilitation (Other)
  Interventions: Behavioral: Modified Constraint-induced Movement Therapy

INTERVENTIONS:
Behavioral: Modified Constraint-induced Movement Therapy — Home based CIT
  1. Restriction of the less affected limb
  2. Intensive practice using affected limb
  3. Positive experience
  4. Functional task (task)
  Other Names: Constraint-Induced Therapy; Forced-use Therapy; Immobilization Therapy

SUMMARY:
This research centers on the comparison of the immediate efficacy (right after therapy) and the maintained efficacy (3 months and 6 months) between "Modified Constraint-Induced Movement Therapy" (mCIMT) group and control group at different age.

DETAILED DESCRIPTION:
"Modified Constraint-Induced Movement Therapy" is one of the most recent treatments for children with Brain damage.

This well-designed and follow-up RCT study compared home-based CIT with a control intervention (traditional rehabilitation, TR) by combining kinematic analysis and clinical evaluation, which is possible to examine whether functional improvement is accompanied by a change in motor control. We hypothesized that home-based CIT would induce better motor control strategies (shorter RT, MT, lesser MUs, MGA, and PMGA, and larger peak velocity (PV)) for greater functional gains than TR. Furthermore, the beneficial effects would be maintained at 3 and 6 months of follow-up. Findings of this study allow clinicians to understand the underlying motor control changes for functional improvement after home-based CIT.

ELIGIBILITY:
Inclusion Criteria:

1. Development learned-nonuse
2. Age range 4y/o-15y/o
3. Wrist ext 10˚, MP j't ext 10˚ in affected U/E
4. Can fallow up the simple instruction
5. Modified Ashworth Scale ≦2
6. Pediatric Motor Activity Log ≦2.5 (average)

Exclusion Criteria:

1. Related muscle skeleton surgery
2. Selective dorsal rhizotomy
3. Botulinum toxin in 6 months
4. Visual perception impaired
5. Hearing perception impaired
6. Balance ability impaired (in constrained)

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Bruininks-Oseretsky Test of Motor Proficiency (BOTMP) | 4 weeks (post-treatment), 12 week, 24 week
  All children underwent a series of upper limb assessments, including kinematic analysis and functional measures (primary and secondary outcomes), before the start of the intervention (pretreatment). An occupational therapist blinded to group assignment was trained to administer these measures. All participants underwent these assessments at 4 weeks immediately after intervention (post-treatment), and at 12-week follow-up and 24-week follow-up.
Peabody Development Motor Scales, subtest fine motor (PDMS-Ⅱ) | 4 weeks (post-treatment), 12 week, 24 week
Kinematic analysis | 4 weeks (post-treatment), 12 week, 24 week

SECONDARY OUTCOMES:
Pediatric Motor Activity Log ( PMAL ) | 4 weeks (post-treatment), 12 week, 24 week
  All children underwent a series of upper limb assessments, including kinematic analysis and functional measures (primary and secondary outcomes), before the start of the intervention (pretreatment). An occupational therapist blinded to group assignment was trained to administer these measures. All participants underwent these assessments at 4 weeks immediately after intervention (post-treatment), and at 12-week follow-up and 24-week follow-up.
Pediatric Functional Independence Measure ( WeeFIM ) | 4 weeks (post-treatment), 12 week, 24 week
Cerebral palsy quality of life (CPQoL) | 4 weeks (post-treatment), 12 week, 24 week

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling chen, MD,PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taoyuan, Taiwan